CLINICAL TRIAL: NCT03416465
Title: Place of General Medical During Oncology Care Management
Acronym: MGPEC_Onco
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A03429-44
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Oncologic Disorders
Keywords: hospitalization; cancer; general practitioner
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: medical questionnaire — The patient will complete a questionnaire of 10 questions before leaving hospital. This questionnaire concerns the care pathway for hospitalized patients.

SUMMARY:
The Purpose of MGPEC_ONCO is to see if patient consult their general practitioner during the management of their cancer, especially before hospitalization. The study concerns not planned hospitalizations in medicine service.

Before leaving hospital, the patient completes the survey, other data are taken in patient record

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing oncology treatment or ≤ 1 year of the latest oncology treatments
* Patient hospitalized in a medical service in an unscheduled way
* Age > or = 18 years old
* Patient informed and not opposed to the study
* Patient able and agreeing to follow all study procédures
* Patient must be affiliated to a social security system

Exclusion Criteria:

* Patient hospitalized in surgery and continuing care services
* Patient deprived of liberty or under supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalized in a medical service in an unscheduled way
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Patients in unscheduled hospitalization | 1 day
  Percentage of patients in unscheduled hospitalization who have seen their general practitioner

CONTACTS AND LOCATIONS:
Overall Officials: HENRY ALINE, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France